CLINICAL TRIAL: NCT05049304
Title: Prevention With Oleanolic Acid of Insulin Resistance and Metabolic Syndrome in Adolescents
Brief Title: Prevention With Oleanolic Acid of Insulin Resistance
Acronym: PREOLIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Emilio Gonzalez Jimenez, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-AGR-287-UGR18
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Insulin Resistance; Metabolic Syndrome
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA-enriched functional olive oil (Experimental)
  Interventions: Other: Functional olive oil
- Olive oil not enriched in OA (Active Comparator)
  Interventions: Other: Olive oil

INTERVENTIONS:
Other: Functional olive oil — Eleven adolescents will consume OA-enriched functional olive oil. After eating the olive oil, aliquots of cubital blood will be drawn at 2 and 5 hours of the postprandial period. During that time, free access to water intake will be allowed.
  Arms: OA-enriched functional olive oil
Other: Olive oil — Eleven adolescents will consume olive oil. After eating the olive oil, aliquots of cubital blood will be drawn at 2 and 5 hours of the postprandial period. During that time, free access to water intake will be allowed.
  Arms: Olive oil not enriched in OA

SUMMARY:
Oleanolic acid (OA), a triterpene that is highly present in olive leaves, has been proposed as component of functional foods in the prevention of metabolic syndrome due to its anti-inflammatory activity. In this research project we will study the presence of OA in postprandial TRL in healthy adolescents and in normal weight. Moreover, THP-1 macrophages will be incubated with LPS for 48h after pretreatment with OA at different concentrations. Also, TRL will be isolated from healthy adolescents before and 2 and 5h postprandially after the intake of a meal containing the functional olive oil or common olive oil and incubated with THP-1 macrophages.

ELIGIBILITY:
Inclusion Criteria:

-Participants without digestive, metabolic or oncologic disorders or any other pathology

Exclusion Criteria:

-Not having the informed consent signed by the parents

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory cytokines | One year
  The pro-inflammatory cytokines were studied in THP-1 macrophages stimulated with postprandial triglyceride-rich lipoproteins

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences (University of Granada), Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided